CLINICAL TRIAL: NCT05124782
Title: Evaluation of Rheumatoid Arthritis at the Time of Telemedicine
Brief Title: Virtual Management of Rheumatoid Arthritis
Acronym: ePRAT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210550
Record Dates: First submitted 2021-10-22; First posted 2021-11-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Virtual consultation; Telemedicine; Patient reported outcome
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with rheumatoid arthritis: Patients seen in virtual consultation
  Interventions: Other: Rheumatoid Arthritis Impact of Disease questionnaire

INTERVENTIONS:
Other: Rheumatoid Arthritis Impact of Disease questionnaire — Rheumatoid Arthritis Impact of Disease questionnaire

SUMMARY:
The purpose of this study is to optimize the care of patients with RA seen in virtual consultation.

DETAILED DESCRIPTION:
This study will be organized in two consecutive steps:

1. A first descriptive step that will consist of a retrospective analysis of virtual consultation records of patients with RA during the pandemic and lockdown period in order to analyze on which criteria the patients were assessed and followed during this period.
2. The second step will consist in evaluating the interest of the systematic use in virtual consultation of a patient reported outcome (PRO), the RAID (Rheumatoid Arthritis Impact of Disease) questionnaire; and analyze how its results influence the rheumatologist decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis fulfilling the 2010 ACR/EULAR classification criteria
* Follow-up in the rheumatology department of Cochin Hospital
* Affiliated with a social security scheme
* Non-opposition to participating in the study
* Patients with a valid email address (registration to the virtual consultation system)

Exclusion Criteria:

* Opposition to participate to this research
* Inability to understand or speak French
* Patient under tutor or curator ship
* patients under medical state help

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatoid arthritis followed in a tertiary center (University Hospital Cochin)
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Rate of face to face consultation, hospitalization and therapeutic modifications | Inclusion
  The primary outcome will be the rate of face to face consultation, hospitalization and therapeutic modifications decided by the rheumatologist during the virtual consultation

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme AVOUAC, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Rheumatology Department, Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No